CLINICAL TRIAL: NCT05115526
Title: Positive End-expiratory Pressure Setting in COVID-19 Related ARDS : Comparison Between Electrical Impedance Tomography, PEEP/ Fraction of Inspired Oxygen Tables, and Transpulmonary Pressure.
Brief Title: PEEP Setting in COVID19-related ARDS
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2021PI117
Record Dates: First submitted 2021-10-15; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: ARDS Due to Severe Acute Respiratory Syndrome Coronavirus 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PEEP setting — PEEP setting according to various methods

SUMMARY:
The best way to titrate positive end-expiratory pressure (PEEP) in patients suffering from acute respiratory distress syndrome is still matter of debate. Electrical impedance tomography (EIT) in a non-invasive technique that could guide PEEP setting based on an optimized ventilation homogeneity.

DETAILED DESCRIPTION:
COVID-19 related ARDS patients admitted to the ICU in March 2021 requiring mechanical ventilation were enrolled. Patients were monitored by an esophageal catheter and a 32-electrode EIT device. Within 48 hours after the start of mechanical ventilation, different levels of PEEP were applied based upon PEEP/ Fraction of inspired oxygen tables, positive end-expiratory transpulmonary (PL)/ FiO2 table, and EIT. Respiratory mechanics variables were recorded.

ELIGIBILITY:
Inclusion Criteria:

* COVID19-related ARDS under invasive mechanical ventilation

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients under mechanical ventilation following COVID19-ARDS
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Value of PEEP | a single determination, within 24-48 hours after mechanical ventilation initiation
  different PEEP values obtained through using different methods

SECONDARY OUTCOMES:
Respiratory mechanics | a single determination, within 24-48 hours after mechanical ventilation initiation
  Respiratory mechanics (plateau pressure, driving pressure, compliance, mechanical power) following different PEEP settings

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Réanimation Médicale, Hôpital Central, Nancy, France

IPD SHARING:
Plan to Share IPD: No